CLINICAL TRIAL: NCT02771652
Title: Effect of an Internet-based At-home Physical Training Protocol on Quality of Life, Fatigue, Functional Performance, Aerobic Capacity and Muscle Strength in Multiple Sclerosis Patients
Acronym: ms-intakt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg (Other)
Collaborators: Caritas-Krankenhaus Bad Mergentheim (Other)
Responsible Party: Principal Investigator, Prof. Dr. Klaus Pfeifer, Prof. Dr., Friedrich-Alexander-Universität Erlangen-Nürnberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.01.1/09/007
Record Dates: First submitted 2016-05-04; First posted 2016-05-13 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Quality of Life; exercise; internet
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- e-training intervention (Active Comparator): Resistance and endurance training
  Interventions: Behavioral: e-training
- Control (Other): no exercise
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: e-training — The e-training intervention is a home-based aerobic and resistance training program. Resistance training was prescribed twice weekly for a period of 12 weeks. No special equipment was necessary except an elastic exercise band or a large gymnastic ball. In addition, endurance training was to be carried out once a week. Training intensity was regulated by the participant's subjective, perceived exertion, which was rated between 6 and 20 on the BORG Scale. The form of activity for the endurance training was freely selected, duration (between 10-60 min) was adjusted to individual fitness levels. Therapists aimed at eliciting a BORG Feedback of between 11 (fairly light) and 16 (hard). The exercise training was home-based and supervised via the internet. Participants continued exercise training for another 12 weeks after the 3month assessment.
  Arms: e-training intervention
Other: Control — After the initial assessment on entry, those assigned to the control group were instructed to maintain their previous physical activity behaviour. After waiting three months, they received the same e-training intervention as the intervention group had received from the start.
  Arms: Control

SUMMARY:
In this randomised controlled trial, the feasibility and effectiveness of an internet-based exercise intervention including progressive strength and endurance training (e-training) for PwMS was investigated. Primary outcome was health-related quality of life, secondary outcomes were muscle strength, aerobic capacity and lung function, physical activity and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed Multiple Sclerosis (McDonald criteria),
* an EDSS score of less than or equal to 4.0,
* not less than 4 weeks of clinical stability prior to inclusion in the study,
* access to the internet.
* the taking of immunotherapeutic agents was not relevant and not monitored

Exclusion Criteria:

* primary progressive multiple sclerosis
* clinically relevant internal disease, especially cardiovascular or pulmonary disease, metabolic and orthopedic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2010-02; Primary Completion 2011-06 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change in Hamburg Quality of Life Questionnaire for Multiple Sclerosis (HAQUAMS) | Assessments took place at baseline and at 3 months
  38 items generate the subscales of fatigue/thinking, mobility of the lower/upper extremities, communication and mood. The HAQUAMS total score is calculated from a mean of the subscales, providing a total score between 1 and 5. Higher scores in HAQUAMS indicate lower levels in HRQoL. The primary outcome will be the change over time from baseline to month 3.

SECONDARY OUTCOMES:
Würzburg Fatigue Scale (WEIMuS) | Assessments took place at baseline, at 3 and 6 months
  This questionnaire contains 17 items that form a physical and cognitive subscale. The total score ranges from zero to a maximum of 68 points (maximum fatigue). The cut-off value for the presence of fatigue is above 32.
Muscle strength lower extremities | Assessments took place at baseline and after 3 and 6 months
  Maximum isometric muscle strength was tested with the M3 Diagnos machine (Schnell, Peutenhausen, Germany).
Forced vital capacity | Assessments took place at baseline and after 3 and 6 months
  Forced vital capacity (FVC) was tested with the Master Screen CPX System (Viasys Healthcare, Cardinal Health, Germany).
Aerobic capacity | Assessments took place at baseline and after 3 and 6 months
  As a marker of endurance capacity, maximal oxygen uptake (VO2peak) was determined by the spiroergometry device Master Screen CPX on a bicycle ergometer (Sanabike 250F, MESA, Germany) at 70-80 revolutions per minute.
Physical activity | Assessments took place at baseline and after 3 and 6 months
  Habitual physical activity was assessed with the German version of the Baecke Questionnaire including three activity indices (work, sport, leisure time PA). There were limitations concerning content validity in all indices; therefore, the sport score of the sport index was used. That score is the product of the intensity, duration and frequency of a participant's reported sports activities. Higher scores indicate a higher level of PA.
Peak expiratory flow | Assessments took place at baseline and after 3 and 6 months
  Peak expiratory flow (PEF) was tested with the Master Screen CPX System (Viasys Healthcare, Cardinal Health, Germany).

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Mäurer, Dr., Principal Investigator — Caritas-Krankenhaus Bad Mergentheim

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tallner A, Tzschoppe R,Peters S, Mäurer M, Pfeifer K. Internetgestützte Bewegungsförderung bei Personen mit Multipler Sklerose. Neurologie und Rehabilitation 19(1): 35-46, 2013.
- Available data/document: Detailed intervention description — https://www.sport.fau.de/files/2016/05/ms-intakt-e-training-intervention-description.pdf — Detailed description of the processes of the e-training intervention (english language)
- Available data/document: Clinical Study Report — https://www.sport.fau.de/files/2015/05/ms-intakt-abschlussbericht-19_05_2015.pdf — Final report for funding foundation (german)